CLINICAL TRIAL: NCT02851108
Title: Safety of Artesunate-amodiaquine Combined With Methylene Blue or Primaquine for Falciparum Malaria Treatment in African Children: A Randomised Controlled Trial
Brief Title: Methylene Blue Against Falciparum Malaria in Burkina Faso
Acronym: BlueACTn
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government)
Responsible Party: Principal Investigator, Olaf Mueller, Prof. Dr., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UniHD008
Record Dates: First submitted 2016-06-28; First posted 2016-08-01 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Malaria, Falciparum
Keywords: falciparum malaria; sub saharan; africa; elimination disorder
MeSH Terms: conditions — Malaria, Falciparum; Elimination Disorders | interventions — Methylene Blue; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AS-AQ-MB (Experimental): Once daily a fixed dose artesunate-amodiaquine formulation combined with once daily methylene blue (15 mg/kg) over a three days period.
  Interventions: Drug: Methylene Blue
- AS-AQ-PQ (Active Comparator): Once daily a fixed dose artesunate-amodiaquine over three days combined with a single dose of primaquine on day 2 (0.25 mg/kg).
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Methylene Blue — 50 patients will receive methylene blue
  Other Names: 3,7-bis(Dimethylamino)-phenothiazine-5-ium chloride
  Arms: AS-AQ-MB
Drug: Primaquine — 50 patients will receive primaquine
  Other Names: (±)-N4-(6-Methoxychinolin-8-yl)pentan-1,4-diamine
  Arms: AS-AQ-PQ

SUMMARY:
Safety of artesunate-amodiaquine combined with methylene blue or primaquine for falciparum malaria treatment in African children: A randomised controlled trial

Elimination has become the goal of malaria programmes in an increasing number of endemic countries and regions. As resistance against artemisinin compounds has recently started to emerge in South-East Asia, there is a clear need to develop alternative malaria drug combinations. Adding another anti-malarial with a short half-life such as methylene blue to standard ACT (artemisinin-based combination therapy) could be a strategy to prevent artemisinin resistance development. Moreover, adding a gametocytocidal drug to ACT reduces the probability of transmission of P. falciparum parasites including drug-resistant parasites.

Objectives: The primary objective of this trial is to investigate the safety of artesunate (AS) - amodiaquine (AQ) - methylene blue (MB) compared to AS - AQ - primaquine (PQ) in young children with uncomplicated falciparum malaria in Burkina Faso.

DETAILED DESCRIPTION:
The overall goal of the underlying research project is to develop a MB-based first-line drug combination regimen against uncomplicated falciparum malaria in SSA.

The primary objective of this study is: To study the safety of the triple combination AS-AQ-MB compared to AS-AQ-PQ in the treatment of uncomplicated falciparum malaria in young African children. The secondary objective of this study is: To study the efficacy of this MB-based triple combination in comparison with standard ACT-PQ in the treatment of uncomplicated falciparum malaria in young African children.

It is a mono-center, open randomised controlled non-inferiority study in children with uncomplicated falciparum malaria in Burkina Faso. Patients will be randomised to two treatment groups (arms):

1. AS-AQ-MB
2. AS-AQ-PQ

Study population: Children aged 6-59 months with uncomplicated falciparum malaria from Nouna Hospital in north-western Burkina Faso.

Sample size: 100 patients (50 per study arm).

Treatment: The group AS-AQ-MB will receive once daily a fixed dose AS-AQ formulation combined with once daily MB (15 mg/kg) over a three days period. The control group will receive once daily a fixed dose AS-AQ over three days combined with a single dose of PQ on day 2 (0.25 mg/kg).

Endpoints: Primary endpoint is the haemoglobin value on day 7 compared to baseline. Secondary endpoints are adverse events (AE), adequate clinical and parasitological response (ACPR) rate (PCR-corrected for recrudescences), as well as gametocyte prevalence and density.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥ 6 kg
* Uncomplicated malaria caused by P. falciparum
* Asexual parasites ≥ 2 000/µl and ≤ 100 000/µl
* Axillary temperature ≥ 37.5°C or a history of fever during the last 24 hours
* Burkinabe nationality
* Permanent residence in the study area with no intention of leaving during the surveillance period
* Written informed consent of parents or care takers

Exclusion Criteria:

* Severe malaria
* Mixed malaria infection
* Vomiting (>2 times within 24 hours before the visit)
* Any apparent significant disease, including severe malnutrition
* A history of a previous, significant adverse reaction or known allergy to one or more of the study drugs
* Anaemia (haemoglobin < 7 g/dl)
* Treated in the same trial before
* All modern antimalarial treatment prior to inclusion (last seven days)
* Therapy with serotonin reuptake inhibitors (e.g. citalopram, escitalopram, fluoxetine, Paroxetine, Sertraline)
* Simultaneous participation in another investigational study
* Patients with known HIV/AIDS disease
* Therapy with drugs known to inhibit the liver enzymes cytochrome 2A6 (e.g. methoxsalen, pilocarpine, tranylcypromine) and/or cytochrome 2C8 (e.g. trimethoprim, ketoconazole, ritonavir, saquinavir, lopinavir, gemfibrozil, montelukast)

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Müller, Prof. Dr., Principal Investigator — Heidelberg University
Locations (1):
- CRSN, Nouna, Burkina Faso

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mendes Jorge M, Ouermi L, Meissner P, Compaore G, Coulibaly B, Nebie E, Krisam J, Klose C, Kieser M, Jahn A, Lu G, D Alessandro U, Sie A, Mockenhaupt FP, Muller O. Safety and efficacy of artesunate-amodiaquine combined with either methylene blue or primaquine in children with falciparum malaria in Burkina Faso: A randomized controlled trial. PLoS One. 2019 Oct 10;14(10):e0222993. doi: 10.1371/journal.pone.0222993. eCollection 2019. PMID 31600221

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AS-AQ-MB | AS-AQ-PQ
Started | 50 | 50
Completed | 42 | 49
Not Completed | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AS-AQ-MB | AS-AQ-PQ | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: months] | 42.34 (12.34) | 38.2 (13.93) | 40.27 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 26 | 25 | 51
Weight [Mean (Standard Deviation); unit: kg] | 12.91 (3.16) | 12.18 (2.98) | 12.55 (3.08)
Length of current disease episode [Mean (Standard Deviation); unit: days] | 1.94 (1.32) | 1.96 (1.28) | 1.95 (1.29)
Prior treatment of current disease episode [Count of Participants; unit: Participants] | 16 | 13 | 29
Any other prior illnesses within last 7 days [Count of Participants; unit: Participants]
  Yes | 4 | 2 | 6
  No | 46 | 48 | 94
Temperature [Mean (Standard Deviation); unit: [°C]] | 37.80 (0.81) | 37.79 (0.79) | 37.80 (0.79)
Hemoglobin [Mean (Standard Deviation); unit: [g/dl]] | 10.16 (1.62) | 9.68 (1.42) | 9.92 (1.53)
P.falciparum merozoites paras. density [Mean (Standard Deviation); unit: parasites/µl blood] | 30373.60 (32808.10) | 23318.80 (25199.72) | 26846.20 (29319.34)
P.falciparum gamotocytes parasite density (for those patients with gametocytes) [Mean (Standard Deviation); unit: parasites/µl blood] | 200.0 (123.29) | 170.0 (110.58) | 181.54 (111.49)
G6PD phenotype [Count of Participants; unit: Participants]
  Deficient | 7 | 7 | 14
  Heterozygous | 11 | 5 | 16
  Normal | 32 | 38 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Haemoglobin Compared to the Baseline
Description: Haemoglobin concentrations will be measured in the field using a HemoCue® (HemoCue® AB, Angelholm, Sweden)
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | AS-AQ-MB | AS-AQ-PQ
Number analyzed (Participants) | 50 | 49
g/dl | 0.18 (1.42) | 0.54 (0.94)

2. Secondary Outcome: Gametocyte Prevalence
Description: measured microscopically at baseline and on day 1, 2, 3, 7, 14, and 28 of follow-up
Time Frame: 28 days
Reporting Status: Not Posted

3. Secondary Outcome: Adverse Events (AE)
Description: Reports of observed or self-reported adverse event
Time Frame: 28 days
Reporting Status: Not Posted

4. Secondary Outcome: Mothers/Caretakers Questionnaire on Acceptance
Description: Acceptance of the different treatment regimens by mothers/caretakers
Time Frame: 14 days
Reporting Status: Not Posted

5. Secondary Outcome: Gametocyte Density
Description: measured microscopically at baseline and on day 1, 2, 3, 7, 14, and 28 of follow-up
Time Frame: 28 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | AS-AQ-MB | AS-AQ-PQ
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/50
Other Adverse Events (participants affected / at risk) | 33/50 | 28/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AS-AQ-MB (N=50) | AS-AQ-PQ (N=50)
Severe anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Severe malaria (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AS-AQ-MB (N=50) | AS-AQ-PQ (N=50)
Gastro-intestinal symptoms (Gastrointestinal disorders) | 14 (19) | 13 (16)
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 20 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No